CLINICAL TRIAL: NCT02397460
Title: A Study to Assess the Effect of AF-219 on Cough Reflex Sensitivity in Both Healthy and Chronic Cough Subjects
Brief Title: Effect of Gefapixant (AF-219/MK-7264) on Cough Reflex Sensitivity (MK-7264-015)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7264-015; AF-219-015 (Other: Afferent Protocol Number); MK-7264-015 (Other: Merck Protocol Number); 2015-000464-34 (EudraCT Number)
Record Dates: First submitted 2015-03-09; First posted 2015-03-25 (Estimated); Results first posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gefapixant 50 mg (Experimental): Gefapixant 50 mg (1 tablet) administered as a single dose
  Interventions: Drug: Gefapixant
- Gefapixant 300 mg (Experimental): Gefapixant 300 mg (6 tablets) administered as a single dose
  Interventions: Drug: Gefapixant
- Placebo (Placebo Comparator): Placebo-matching tablets administered as a single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gefapixant — Gefapixant tablets administered orally as a single dose of 50 mg (1 tablet) or 300 mg (6 tablets)
  Other Names: AF-219; MK-7264
  Arms: Gefapixant 300 mg; Gefapixant 50 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this double-blind crossover study is to assess the effect of single doses of 50 mg and 300 mg gefapixant (AF-219/MK-7264) on cough reflex sensitivity to capsaicin in both healthy participants and participants with chronic cough. This study will also assess the effect of single doses of gefapixant on cough reflex sensitivity to adenosine triphosphate (ATP) in healthy participants and participants with chronic cough.

DETAILED DESCRIPTION:
Up to 30 participants (male and female) who meet all entry criteria will be randomly assigned to treatment with gefapixant or matching placebo.

There will be a Screening Period, a Baseline Visit (cough participants only), and four Treatment Periods, with a washout period between treatments. Participants will return after their last Treatment Visit for a Follow-up Visit.

At the Screening Visit and during the Treatment Periods, cough sensitivity will be measured by standard clinical methodology incorporating two cough challenges: 1) capsaicin; 2) ATP. The ATP challenge will only be performed during the study treatment period. The Baseline Visit (cough participants only) will occur prior to Treatment Period 1. Daytime cough monitoring will be performed at the Baseline Visit and during each of the four Treatment Periods (cough participants only).

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed voluntary consent;
* Be able to speak, read, and understand English;
* Be males or females, of any race, between 18 and 80 years of age, inclusive;
* Have a body mass index (BMI) ≥18 and <35.0 kg/m2;
* Be in good general health with no clinically relevant abnormalities based on the medical history, physical examination, clinical laboratory evaluations (hematology, clinical chemistry, and urinalysis), and 12 lead electrocardiogram;
* Women of child bearing potential must have a negative pregnancy test at Screening and prior to randomization.
* Women of child-bearing potential must use 2 methods of acceptable birth control from Screening until 3 months after the last dose of study drug;
* Male subjects with partners of child-bearing potential (as defined in Inclusion No. 8) must use 2 methods of acceptable birth control, 1 of which must be a barrier method;
* Subjects with chronic cough
* Be able to communicate effectively with the Investigator and other study center personnel and agree to comply with the study procedures and restrictions

Exclusion Criteria:

* Current smoker;
* Individuals who have given up smoking within the past 6 months, or those with >20 pack-year smoking history(chronic cough subjects), or >10 pack-year smoking history (healthy subjects);
* History of upper respiratory tract infection or recent significant change in pulmonary status within 4 weeks prior to Screening or prior to randomization;
* History of concurrent malignancy or recurrence of malignancy within 2 years prior to Screening (with the exception of < 3 excised basal cell carcinomas);
* History of a diagnosis of drug or alcohol dependency or abuse within the last 3 years;
* In the opinion of the Principal Investigator, an uncontrolled or unstable clinically significant neurological, psychiatric, respiratory, cardiovascular, peripheral vascular, gastrointestinal, hepatic, pancreatic, endocrinological, hematological, or immunological disorder or an active infection;
* Clinically significant abnormal electrocardiogram (ECG) at Screening
* Significantly abnormal laboratory tests at Screening
* Breastfeeding;
* In the judgement of the Principal Investigator, other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and would make the subject inappropriate for entry into this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- The Medicines Evaluation Unit, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: PBO→Gefapixant 300 mg→PBO→Gefapixant 300 mg/Healthy: Healthy participants in Cohort 1/Sequence A received single doses of placebo (PBO) on Day 1 of Periods 1 and 3 and single doses of gefapixant 300 mg on Day 1 of Periods 2 and 4. (Each treatment period consisted of Day 1 and Day 2.) There was a minimum 48-hour washout period between treatment periods.
- Cohort 1: Gefapixant 300 mg→PBO→Gefapixant 300 mg→PBO/Healthy: Healthy participants in Cohort 1/Sequence B received single doses of gefapixant 300 mg on Day 1 of Periods 1 and 3 and singles doses of placebo on Day 1 of Periods 2 and 4. (Each treatment period consisted of Day 1 and Day 2.) There was a minimum 48-hour washout period between treatment periods.
- Cohort 1: PBO→Gefapixant 300 mg→PBO→Gefapixant 300 mg/CC: Participants with chronic cough (CC) in Cohort 1/Sequence A received singles doses of placebo on Day 1 of Periods 1 and 3 and single doses of gefapixant 300 mg on Day 1 of Periods 2 and 4. (Each treatment period consisted of Day 1 and Day 2.) There was a minimum 48-hour washout period between treatment periods.
- Cohort 1: Gefapixant 300 mg→PBO→Gefapixant 300 mg→PBO/CC: Participants with chronic cough in Cohort 1/Sequence B received singles doses of gefapixant 300 mg on Day 1 of Periods 1 and 3 and single doses of placebo on Day 1 of Periods 2 and 4. (Each treatment period consisted of Day 1 and Day 2.) There was a minimum 48-hour washout period between treatment periods.
- Cohort 2: PBO→Gefapixant 50 mg→PBO→Gefapixant 50 mg/Healthy: Healthy participants in Cohort 2/Sequence A received singles doses of placebo on Day 1 of Periods 1 and 3 and single doses of gefapixant 50 mg on Day 1 of Periods 2 and 4. (Each treatment period consisted of Day 1 and Day 2.) There was a minimum 48-hour washout period between treatment periods.
- Cohort 2: Gefapixant 50 mg→PBO→Gefapixant 50 mg→PBO/Healthy: Healthy participants in Cohort 2/Sequence B received single doses of gefapixant 50 mg on Day 1 of Periods 1 and 3 and single doses of placebo on Day 1 of Periods 2 and 4. (Each treatment period consisted of Day 1 and Day 2.) There was a minimum 48-hour washout period between treatment periods.
- Cohort 2: PBO→Gefapixant 50 mg→PBO→Gefapixant 50 mg/CC: Participants with chronic cough in Cohort 2/Sequence A received singles doses of placebo on Day of Periods 1 and 3 and singles doses of gefapixant 50 mg on Day 1 of Periods 2 and 4. (Each treatment period consisted of Day 1 and Day 2.) There was a minimum 48-hour washout period between treatment periods.
- Cohort 2: Gefapixant 50 mg→PBO→Gefapixant 50 mg→PBO/CC: Participants with chronic cough in Cohort 2/Sequence B received singles doses of gefapixant 50 mg on Day 1 of Periods 1 and 3 and singles doses of placebo on Day 1 of Periods 2 and 4. (Each treatment period consisted of Day 1 and Day 2.) There was a minimum 48-hour washout period between treatment periods.
Period: Treatment Period 1
Arm/Group | Cohort 1: PBO→Gefapixant 300 mg→PBO→Gefapixant 300 mg/Healthy | Cohort 1: Gefapixant 300 mg→PBO→Gefapixant 300 mg→PBO/Healthy | Cohort 1: PBO→Gefapixant 300 mg→PBO→Gefapixant 300 mg/CC | Cohort 1: Gefapixant 300 mg→PBO→Gefapixant 300 mg→PBO/CC | Cohort 2: PBO→Gefapixant 50 mg→PBO→Gefapixant 50 mg/Healthy | Cohort 2: Gefapixant 50 mg→PBO→Gefapixant 50 mg→PBO/Healthy | Cohort 2: PBO→Gefapixant 50 mg→PBO→Gefapixant 50 mg/CC | Cohort 2: Gefapixant 50 mg→PBO→Gefapixant 50 mg→PBO/CC
Started | 7 | 7 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 7 | 7 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Cohort 1: PBO→Gefapixant 300 mg→PBO→Gefapixant 300 mg/Healthy | Cohort 1: Gefapixant 300 mg→PBO→Gefapixant 300 mg→PBO/Healthy | Cohort 1: PBO→Gefapixant 300 mg→PBO→Gefapixant 300 mg/CC | Cohort 1: Gefapixant 300 mg→PBO→Gefapixant 300 mg→PBO/CC | Cohort 2: PBO→Gefapixant 50 mg→PBO→Gefapixant 50 mg/Healthy | Cohort 2: Gefapixant 50 mg→PBO→Gefapixant 50 mg→PBO/Healthy | Cohort 2: PBO→Gefapixant 50 mg→PBO→Gefapixant 50 mg/CC | Cohort 2: Gefapixant 50 mg→PBO→Gefapixant 50 mg→PBO/CC
Started | 7 | 7 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 7 | 7 | 6 | 6 | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 3
Arm/Group | Cohort 1: PBO→Gefapixant 300 mg→PBO→Gefapixant 300 mg/Healthy | Cohort 1: Gefapixant 300 mg→PBO→Gefapixant 300 mg→PBO/Healthy | Cohort 1: PBO→Gefapixant 300 mg→PBO→Gefapixant 300 mg/CC | Cohort 1: Gefapixant 300 mg→PBO→Gefapixant 300 mg→PBO/CC | Cohort 2: PBO→Gefapixant 50 mg→PBO→Gefapixant 50 mg/Healthy | Cohort 2: Gefapixant 50 mg→PBO→Gefapixant 50 mg→PBO/Healthy | Cohort 2: PBO→Gefapixant 50 mg→PBO→Gefapixant 50 mg/CC | Cohort 2: Gefapixant 50 mg→PBO→Gefapixant 50 mg→PBO/CC
Started | 7 | 7 | 6 | 6 | 6 | 6 | 6 | 5
Completed | 7 | 7 | 6 | 6 | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Cohort 1: PBO→Gefapixant 300 mg→PBO→Gefapixant 300 mg/Healthy | Cohort 1: Gefapixant 300 mg→PBO→Gefapixant 300 mg→PBO/Healthy | Cohort 1: PBO→Gefapixant 300 mg→PBO→Gefapixant 300 mg/CC | Cohort 1: Gefapixant 300 mg→PBO→Gefapixant 300 mg→PBO/CC | Cohort 2: PBO→Gefapixant 50 mg→PBO→Gefapixant 50 mg/Healthy | Cohort 2: Gefapixant 50 mg→PBO→Gefapixant 50 mg→PBO/Healthy | Cohort 2: PBO→Gefapixant 50 mg→PBO→Gefapixant 50 mg/CC | Cohort 2: Gefapixant 50 mg→PBO→Gefapixant 50 mg→PBO/CC
Started | 7 | 7 | 6 | 6 | 6 | 6 | 6 | 5
Completed | 7 | 6 | 6 | 6 | 5 | 6 | 6 | 5
Not Completed | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: PBO→Gefapixant 300 mg→PBO→Gefapixant 300 mg/Healthy | Cohort 1: Gefapixant 300 mg→PBO→Gefapixant 300 mg→PBO/Healthy | Cohort 1: PBO→Gefapixant 300 mg→PBO→Gefapixant 300 mg/CC | Cohort 1: Gefapixant 300 mg→PBO→Gefapixant 300 mg→PBO/CC | Cohort 2: PBO→Gefapixant 50 mg→PBO→Gefapixant 50 mg/Healthy | Cohort 2: Gefapixant 50 mg→PBO→Gefapixant 50 mg→PBO/Healthy | Cohort 2: PBO→Gefapixant 50 mg→PBO→Gefapixant 50 mg/CC | Cohort 2: Gefapixant 50 mg→PBO→Gefapixant 50 mg→PBO/CC | Total
Number analyzed (Participants) | 7 | 7 | 6 | 6 | 6 | 6 | 6 | 6 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.1 (11.87) | 40.9 (6.20) | 61.0 (9.25) | 59.5 (8.38) | 35.0 (8.17) | 34.7 (7.42) | 60.5 (6.83) | 55 (9.01) | 47.2 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 5 | 5 | 0 | 0 | 5 | 4 | 19
  Male | 7 | 7 | 1 | 1 | 6 | 6 | 1 | 2 | 31

OUTCOME MEASURES:

1. Primary Outcome: Cough Reflex Sensitivity to Capsaicin Measured by Maximal Cough Response (Emax)
Description: The effect of single doses of 50 mg and 300 mg gefapixant on cough reflex sensitivity to challenge with capsaicin was assessed in male and female healthy participants and participants with chronic cough. Capsaicin-evoked cough challenge was performed 2 hours post-dose in Periods 1 and 2. The maximal cough response (Emax) to capsaicin was assessed. For capsaicin challenge, doubling concentrations from 0.49 μM to 1000 μM were prepared by dilution of stock solutions with saline, and were administered by inhalation. The number of explosive cough sounds occurring within the first 15 seconds after inhalation were recorded. Nonlinear mixed-effects modeling was used to estimate the Emax. Population pharmacodynamic modeling was performed in NONMEM 7.3. Data exploration, goodness-of-fit plots, statistical analyses, and simulations were performed in Matlab R2015a. Note: All values presented in this table are model-based.
Time Frame: 2 hours post-dose
Population: All randomized participants who received at least 1 dose of study medication and had at least 1 post-dose primary endpoint assessment of Emax in response to capsaicin challenge
Measure: Number; unit: Emax (Explosive coughs/15 sec)
Groups:
- Placebo/Healthy Males: Healthy males who received single doses of placebo in Periods 1 and 2
- Placebo/Chronic Cough Males: Males with chronic cough who received single doses of placebo in Periods 1 and 2
- Placebo/Chronic Cough Females: Females with chronic cough who received single doses of placebo in Periods 1 and 2
- Gefapixant 50 mg/Healthy Males: Healthy males who received single doses of gefapixant 50 mg in Periods 1 and 2
- Gefapixant 50 mg/Chronic Cough Males: Males with chronic cough who received single doses of gefapixant 50 mg in Periods 1 and 2
- Gefapixant 50 mg/Chronic Cough Females: Females with chronic cough who received single doses of gefapixant 50 mg in Periods 1 and 2
- Gefapixant 300 mg/Healthy Males: Healthy males who received single doses of gefapixant 300 mg in Periods 1 and 2
- Gefapixant 300 mg/Chronic Cough Males: Males with chronic cough who received single doses of gefapixant 300 mg in Periods 1 and 2
- Gefapixant 300 mg/Chronic Cough Females: Females with chronic cough who received single doses of gefapixant 300 mg in Periods 1 and 2
Arm/Group | Placebo/Healthy Males | Placebo/Chronic Cough Males | Placebo/Chronic Cough Females | Gefapixant 50 mg/Healthy Males | Gefapixant 50 mg/Chronic Cough Males | Gefapixant 50 mg/Chronic Cough Females | Gefapixant 300 mg/Healthy Males | Gefapixant 300 mg/Chronic Cough Males | Gefapixant 300 mg/Chronic Cough Females
Number analyzed (Participants) | 26 | 5 | 18 | 26 | 5 | 18 | 26 | 5 | 18
Emax (Explosive coughs/15 sec) | 4.14 | 4.14 | 7.57 | 3.66 | 3.37 | 6.17 | 3.66 | 3.37 | 6.17
Statistical Analysis 1: Comparison: Placebo/Healthy Males vs Placebo/Chronic Cough Males vs Placebo/Chronic Cough Females vs Gefapixant 50 mg/Healthy Males vs Gefapixant 50 mg/Chronic Cough Males vs Gefapixant 50 mg/Chronic Cough Females vs Gefapixant 300 mg/Healthy Males vs Gefapixant 300 mg/Chronic Cough Males vs Gefapixant 300 mg/Chronic Cough Females; Treatment effects on Emax following capsaicin challenge were modeled for dose dependence and were estimated on the basis of disease status for participants who were healthy or had chronic cough and received gefapixant 50 mg, gefapixant 300 mg, or placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

2. Primary Outcome: Cough Reflex Sensitivity to Capsaicin Measured by the Tussive Concentration Required to Achieve 50% of Emax (ED50)
Description: The effect of single doses of 50 mg and 300 mg gefapixant on cough reflex sensitivity to challenge with capsaicin was assessed in male and female healthy participants and participants with chronic cough. Capsaicin-evoked cough challenge was performed 2 hours post-dose in Periods 1 and 2. The concentration of capsaicin required to induce 50% of the Emax (ED50) was assessed. For capsaicin challenge, doubling concentrations from 0.49 μM to 1000 μM were prepared by dilution of stock solutions with saline, and were administered by inhalation. Nonlinear mixed-effects modeling was used to estimate the ED50. Population pharmacodynamic modeling was performed in NONMEM 7.3 using Laplace estimation method. Data exploration, goodness-of-fit plots, statistical analyses, and simulations were performed in Matlab R2015a. Note: All values presented in this table are model-based.
Time Frame: 2 hours post-dose
Population: All randomized participants who received at least 1 dose of study medication and had at least 1 post-dose primary endpoint assessment of ED50 in response to capsaicin challenge
Measure: Number; unit: µM
Arm/Group | Placebo/Healthy Males | Placebo/Chronic Cough Males | Placebo/Chronic Cough Females | Gefapixant 50 mg/Healthy Males | Gefapixant 50 mg/Chronic Cough Males | Gefapixant 50 mg/Chronic Cough Females | Gefapixant 300 mg/Healthy Males | Gefapixant 300 mg/Chronic Cough Males | Gefapixant 300 mg/Chronic Cough Females
Number analyzed (Participants) | 26 | 5 | 18 | 26 | 5 | 18 | 26 | 5 | 18
µM | 33 | 33 | 9.56 | 33 | 33 | 9.56 | 33 | 33 | 9.56
Statistical Analysis 1: Comparison: Placebo/Healthy Males vs Placebo/Chronic Cough Males vs Placebo/Chronic Cough Females vs Gefapixant 50 mg/Healthy Males vs Gefapixant 50 mg/Chronic Cough Males vs Gefapixant 50 mg/Chronic Cough Females vs Gefapixant 300 mg/Healthy Males vs Gefapixant 300 mg/Chronic Cough Males vs Gefapixant 300 mg/Chronic Cough Females; Treatment effects following capsaicin challenge were modeled for dose. dependence and were estimated on the basis of disease status for participants who had chronic cough and received gefapixant 50 mg, gefapixant 300 mg, or placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis

3. Secondary Outcome: Cough Reflex Sensitivity to Adenosine Triphosphate (ATP) Measured by Maximal Cough Response (Emax)
Description: The effect of single doses of 50 mg and 300 mg gefapixant on cough reflex sensitivity to challenge with adenosine triphosphate (ATP) was assessed in male and female healthy participants and participants with chronic cough. ATP-evoked cough challenge was performed 2 hours post-dose in Periods 3 and 4. For ATP challenge, doubling concentrations from 0.227 μmol/mL to 929 μmol/mL were prepared from ATP powder dissolved in saline, and were administered by inhalation. The number of explosive cough sounds occurring within the first 15 seconds after inhalation were recorded. Nonlinear mixed-effects modeling was used to estimate the Emax. Population pharmacodynamic modeling was performed in NONMEM 7.3. Data exploration, goodness-of-fit plots, statistical analyses, and simulations were performed in Matlab R2015a. Note: All values presented in this table are model-based.
Time Frame: 2 hours post-dose
Population: All randomized participants who received at least 1 dose of study medication and had at least 1 post-dose secondary endpoint assessment of Emax in response to ATP challenge
Measure: Number; unit: Emax (Explosive coughs/15 sec)
Groups:
- Placebo/Healthy Males: Healthy males who received single doses of placebo in Periods 3 and 4
- Placebo/Chronic Cough Males: Chronic cough males who received single doses of placebo in Periods 3 and 4
- Placebo/Chronic Cough Females: Females with chronic cough who received single doses of placebo in Periods 3 and 4
- Gefapixant 50 mg/Healthy Males: Healthy males who received single doses of gefapixant 50 mg in Periods 3 and 4
- Gefapixant 50 mg/Chronic Cough Males: Males with chronic cough who received single doses of gefapixant 50 mg in Periods 3 and 4
- Gefapixant 50 mg/Chronic Cough Females: Females with chronic cough who received single doses of gefapixant 50 mg in Periods 3 and 4
- Gefapixant 300 mg/Healthy Males: Healthy males who received single doses of gefapixant 300 mg in Periods 3 and 4
- Gefapixant 300 mg/Chronic Cough Males: Males with chronic cough who received single doses of gefapixant 300 mg in Periods 3 and 4
- Gefapixant 300 mg/Chronic Cough Females: Females with chronic cough who received single doses of gefapixant 300 mg in Periods 3 and 4
Arm/Group | Placebo/Healthy Males | Placebo/Chronic Cough Males | Placebo/Chronic Cough Females | Gefapixant 50 mg/Healthy Males | Gefapixant 50 mg/Chronic Cough Males | Gefapixant 50 mg/Chronic Cough Females | Gefapixant 300 mg/Healthy Males | Gefapixant 300 mg/Chronic Cough Males | Gefapixant 300 mg/Chronic Cough Females
Number analyzed (Participants) | 26 | 4 | 18 | 26 | 4 | 18 | 26 | 4 | 18
Emax (Explosive coughs/15 sec) | 2.35 | 2.35 | 5.4 | 2.35 | 2.35 | 5.4 | 2.35 | 2.35 | 5.4

4. Secondary Outcome: Cough Reflex Sensitivity to ATP Measured by the Tussive Concentration Required to Achieve 50% of Emax (ED50)
Description: The effect of single doses of 50 mg and 300 mg gefapixant on cough reflex sensitivity to challenge with ATP was assessed in male and female healthy participants and participants with chronic cough. ATP-evoked cough challenge was performed 2 hours post-dose in Periods 3 and 4. The concentration of ATP required to induce 50% of the Emax (ED50) was assessed. For ATP challenge, doubling concentrations from 0.227 μmol/mL to 929 μmol/mL were prepared by dilution of stock solutions with saline, and were administered by inhalation. Nonlinear mixed-effects modeling was used to estimate the ED50. Population pharmacodynamic modeling was performed in NONMEM 7.3 using Laplace estimation method. Data exploration, goodness-of-fit plots, statistical analyses, and simulations were performed in Matlab R2015a. Note: All values presented in this table are model-based.
Time Frame: 2 hours post-dose
Population: All randomized participants who received at least 1 dose of study medication and had at least 1 post-dose secondary endpoint assessment of ED50 in response to ATP challenge
Measure: Number; unit: µmol/mL
Arm/Group | Placebo/Healthy Males | Placebo/Chronic Cough Males | Placebo/Chronic Cough Females | Gefapixant 50 mg/Healthy Males | Gefapixant 50 mg/Chronic Cough Males | Gefapixant 50 mg/Chronic Cough Females | Gefapixant 300 mg/Healthy Males | Gefapixant 300 mg/Chronic Cough Males | Gefapixant 300 mg/Chronic Cough Females
Number analyzed (Participants) | 14 | 4 | 18 | 26 | 4 | 18 | 26 | 4 | 18
µmol/mL | 54.9 | 54.9 | 8.63 | 119.13 | 155.92 | 24.51 | 119.13 | 192.7 | 30.29

5. Secondary Outcome: Concentrations of Capsaicin Inducing 2 or More Coughs (C2)
Description: The concentrations of capsaicin inducing 2 or more coughs (C2) in participants were assessed in Periods 1 and 2. For capsaicin challenge, doubling concentrations from 0.49 μM to 1000 μM were prepared by dilution of stock solutions with saline, and were administered by inhalation.
Time Frame: 2 hours post-dose
Population: All randomized participants who received at least 1 dose of study medication and had at least 1 post-dose secondary endpoint assessment of C2 in response to capsaicin challenge
Measure: Median (Full Range); unit: µM
Groups:
- Cohort 1: Gefapixant 300 mg/Healthy: Healthy males and females in Cohort 1 who received single doses of gefapixant 300 mg in Periods 1 and 2 combined
- Cohort 1: Placebo/Healthy: Healthy males and females in Cohort 1 who received single doses of placebo in Periods 1 and 2 combined
- Cohort 1: Gefapixant 300 mg/Chronic Cough: Males and females with chronic cough in Cohort 1 who received single doses of gefapixant 300 mg in Periods 1 and 2 combined
- Cohort 1: Placebo/Chronic Cough: Males and females in Cohort 1 with chronic cough who received single doses of placebo in Periods 1 and 2 combined
- Cohort 2: Gefapixant 50 mg/Healthy: Healthy males and females who received single doses of gefapixant 50 mg in Periods 1 and 2 combined
- Cohort 2: Placebo/Healthy: Healthy males and females in Cohort 2 who received single doses of placebo in Periods 1 and 2 combined
- Cohort 2: Gefapixant 50 mg/Chronic Cough: Males and females with chronic cough in Cohort 2 who received single doses of gefapixant 50 mg in Periods 1 and 2 combined
- Cohort 2: Placebo/Chronic Cough: Males and females with chronic cough in Cohort 2 who received single doses of placebo in Periods 1 and 2 combined
Arm/Group | Cohort 1: Gefapixant 300 mg/Healthy | Cohort 1: Placebo/Healthy | Cohort 1: Gefapixant 300 mg/Chronic Cough | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Healthy | Cohort 2: Placebo/Healthy | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 14 | 10 | 10 | 12 | 12 | 10 | 12
µM | 31.25 [4 to 1000] | 31.25 [4 to 500] | 3.90 [0 to 16] | 7.81 [0 to 31] | 15.62 [2 to 63] | 23.44 [8 to 125] | 15.62 [0 to 125] | 5.86 [0 to 250]

6. Secondary Outcome: Concentrations of Capsaicin Inducing 5 or More Coughs (C5)
Description: The concentrations of capsaicin inducing 5 or more coughs (C5) in participants were assessed in Periods 1 and 2. For capsaicin challenge, doubling concentrations from 0.49 μM to 1000 μM were prepared by dilution of stock solutions with saline, and were administered by inhalation.
Time Frame: 2 hours post-dose
Population: All randomized participants who received at least 1 dose of study medication and had at least 1 post-dose secondary endpoint assessment of C5 in response to capsaicin challenge
Measure: Median (Full Range); unit: µM
Groups:
- Cohort 1: Placebo/Chronic Cough: Males and females with chronic cough in Cohort 1 who received single doses of placebo in Periods 1 and 2 combined
- Cohort 2: Gefapixant 50 mg/Healthy: Healthy males and females in Cohort 2 who received single doses of gefapixant 50 mg in Periods 1 and 2 combined
Arm/Group | Cohort 1: Gefapixant 300 mg/Healthy | Cohort 1: Placebo/Healthy | Cohort 1: Gefapixant 300 mg/Chronic Cough | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Healthy | Cohort 2: Placebo/Healthy | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
Number analyzed (Participants) | 5 | 6 | 10 | 10 | 6 | 7 | 7 | 10
µM | 31.25 [16 to 250] | 62.50 [16 to 1000] | 3.90 [0 to 31] | 11.72 [0 to 125] | 250.00 [63 to 500] | 125.00 [63 to 500] | 15.62 [2 to 63] | 5.86 [0 to 31]

7. Secondary Outcome: Concentrations of ATP Inducing 2 or More Coughs (C2)
Description: The concentrations of ATP inducing 2 or more coughs (C2) in participants were assessed in Periods 3 and 4. For ATP challenge, doubling concentrations from 0.227 to 929 μmol/mL were prepared from ATP powder, dissolved and diluted in saline, and administered by inhalation.
Time Frame: 2 hours post-dose
Population: All randomized participants who received at least 1 dose of study medication and had at least 1 post-dose secondary endpoint assessment of C2 in response to ATP challenge
Measure: Median (Full Range); unit: mg/mL
Groups:
- Cohort 1: Gefapixant 300 mg/Healthy: Healthy males and females in Cohort 1 who received single doses of gefapixant 300 mg in Periods 3 and 4 combined
- Cohort 1: Placebo/Healthy: Healthy males and females in Cohort 1 who received single doses of placebo in Periods 3 and 4 combined
- Cohort 1: Gefapixant 300 mg/Chronic Cough: Males and females with chronic cough in Cohort 1 who received single doses of gefapixant 300 mg in Periods 3 and 4 combined
- Cohort 1: Placebo/Chronic Cough: Males and females with chronic cough in Cohort 1 who received single doses of placebo in Periods 3 and 4 combined
- Cohort 2: Gefapixant 50 mg/Healthy: Healthy males and females in Cohort 2 who received single doses of gefapixant 50 mg in Periods 3 and 4 combined
- Cohort 2: Placebo/Healthy: Healthy males and females in Cohort 2 who received single doses of placebo in Periods 3 and 4 combined
- Cohort 2: Gefapixant 50 mg/Chronic Cough: Males and females with chronic cough in Cohort 2 who received single doses of gefapixant 50 mg in Periods 3 and 4 combined
- Cohort 2: Placebo/Chronic Cough: Males and females with chronic cough in Cohort 2 who received single doses of placebo in Periods 3 and 4 combined
Arm/Group | Cohort 1: Gefapixant 300 mg/Healthy | Cohort 1: Placebo/Healthy | Cohort 1: Gefapixant 300 mg/Chronic Cough | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Healthy | Cohort 2: Placebo/Healthy | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
Number analyzed (Participants) | 10 | 11 | 7 | 11 | 9 | 8 | 8 | 9
mg/mL | 192.00 [8 to 256] | 64.00 [1 to 512] | 8.00 [0 to 64] | 1.00 [0 to 64] | 16.00 [8 to 256] | 24.00 [2 to 512] | 4.25 [0 to 512] | 4.00 [0 to 256]

8. Secondary Outcome: Concentrations of ATP Inducing 5 or More Coughs (C5)
Description: The concentrations of ATP inducing 5 or more coughs (C5) in participants were assessed in Periods 3 and 4. For ATP challenge, doubling concentrations from 0.227 to 929 μmol/mL were prepared from ATP powder, dissolved and diluted in saline, and administered by inhalation.
Time Frame: 2 hours post-dose
Population: All randomized participants who received at least 1 dose of study medication and had at least 1 post-dose secondary endpoint assessment of C5 in response to ATP challenge
Measure: Median (Full Range); unit: mg/mL
Groups:
- Cohort 1: Chronic Cough/Gefapixant 300 mg: Males and females with chronic cough in Cohort 1 who received single doses of gefapixant 300 mg in Periods 3 and 4 combined
- Cohort 2: Placebo/Chronic Cough: Males and females with chronic cough in Cohort 2 who received placebo in Periods 3 and 4 combined
Arm/Group | Cohort 1: Gefapixant 300 mg/Healthy | Cohort 1: Placebo/Healthy | Cohort 1: Chronic Cough/Gefapixant 300 mg | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Healthy | Cohort 2: Placebo/Healthy | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
Number analyzed (Participants) | 2 | 5 | 7 | 8 | 4 | 4 | 5 | 8
mg/mL | 192.00 [128 to 256] | 128.00 [64 to 256] | 8.00 [0 to 64] | 16.50 [0 to 512] | 64.00 [32 to 256] | 32.00 [2 to 32] | 128.00 [8 to 512] | 4.00 [0 to 128]

9. Secondary Outcome: Urge-to-Cough in Response to Capsaicin Challenge (Chronic Cough Participants Only)
Description: In response to capsaicin challenges in Periods 1 and 2, participants with chronic cough completed a visual analogue scale (VAS) at the end of a 4-hour post-dose observation period on Day 1; and at end of 24-hour observation period on Day 2. For both periods, participants were asked to mark on a 100 mm VAS the severity of their urge to cough between 0 mm (no urge-to-cough) and 100 mm (worst urge-to-cough).
Time Frame: At the end of a 4-hour post-dose observation period on Day 1; at the end of a 24-hour observation period on Day 2
Population: All randomized participants with chronic cough who received at least 1 dose of study medication and had at least 1 post-dose secondary endpoint assessment of urge-to-cough in response to capsaicin challenge
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Cohort 1: Gefapixant 300 mg/Chronic Cough: Participants with chronic cough in Cohort 1 who received single doses of gefapixant 300 mg in Periods 1 and 2 combined
- Cohort 1: Placebo/Chronic Cough: Participants with chronic cough in Cohort 1 who received single doses of placebo in Periods 1 and 2 combined
- Cohort 2: Gefapixant 50 mg/Chronic Cough: Participants with chronic cough in Cohort 2 who received single doses of gefapixant 50 mg in Periods 1 and 2 combined
- Cohort 2: Placebo/Chronic Cough: Participants with chronic cough in Cohort 2 who received single doses of placebo in Periods 1 and 2 combined
Arm/Group | Cohort 1: Gefapixant 300 mg/Chronic Cough | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 12 | 12 | 11
Score on a scale
  Day 1 | 28.9 (29.79) | 38.6 (26.82) | 36.6 (30.84) | 20.5 (11.54)
  Day 2 | 28.2 (32.72) | 46.7 (29.20) | 41.8 (31.02) | 36.7 (23.28)

10. Secondary Outcome: Urge-to-Cough in Response to ATP Challenge (Chronic Cough Participants Only)
Description: In response to ATP challenges in Periods 3 and 4, participants with chronic cough completed a VAS at the end of a 4-hour post-dose observation period on Day 1; and at end of 24-hour observation period on Day 2. For both periods, participants were asked to mark on a 100 mm VAS the severity of their urge to cough between 0 mm (no urge-to-cough) and 100 mm (worst urge-to-cough).
Time Frame: At the end of a 4-hour post-dose observation period on Day 1; at the end of a 24-hour observation period on Day 2
Population: All randomized participants with chronic cough who received at least 1 dose of study medication and had at least 1 post-dose secondary endpoint assessment of urge-to-cough in response to ATP challenge
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Cohort 1: Gefapixant 300 mg/Chronic Cough: Participants with chronic cough in Cohort 1 who received single doses of gefapixant 300 mg in Periods 3 and 4 combined
- Cohort 1: Placebo/Chronic Cough: Participants with chronic cough in Cohort 1 who received single doses of placebo in Periods 3 and 4 combined
- Cohort 2: Gefapixant 50 mg/Chronic Cough: Participants with chronic cough in Cohort 2 who received single doses of gefapixant 50 mg in Periods 3 and 4 combined
- Cohort 2: Placebo/Chronic Cough: Participants with chronic cough in Cohort 2 who received single doses of placebo in Periods 3 and 4 combined
Arm/Group | Cohort 1: Gefapixant 300 mg/Chronic Cough | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 12 | 11 | 11
Score on a scale
  Day 1 | 19.8 (23.54) | 34.4 (26.78) | 21.5 (22.45) | 25.3 (19.69)
  Day 2 | 21.6 (20.65) | 39.8 (26.51) | 27.5 (29.54) | 37.5 (27.33)

11. Secondary Outcome: Cough Severity in Response to Capsaicin Challenge (Chronic Cough Participants Only)
Description: In response to capsaicin challenges in Periods 1 and 2, participants with chronic cough completed a VAS at the end of a 4-hour post-dose observation period on Day 1; and at end of 24-hour observation period on Day 2. For both periods, participants were asked to mark on a 100 mm VAS their cough severity between 0 mm (no cough) and 100 mm (worst cough).
Time Frame: At the end of a 4-hour post-dose observation period; at the end of a 24-hour observation period on Day 2
Population: All randomized participants with chronic cough who received at least 1 dose of study medication and had at least 1 post-dose secondary endpoint assessment of cough severity in response to capsaicin challenge
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Cohort 1: Gefapixant 300 mg/Chronic Cough: Participants with chronic cough in Cohort 1 who received gefapixant 300 mg in Periods 1 and 2 combined
- Cohort 1: Placebo/Chronic Cough: Participants with chronic cough in Cohort 1 who received placebo in Periods 1 and 2 combined
- Cohort 2: Gefapixant 50 mg/Chronic Cough: Participants with chronic cough in Cohort 2 who received gefapixant 50 mg in Periods 1 and 2 combined
- Cohort 2: Placebo/Chronic Cough: Participants with chronic cough in Cohort 2 who received placebo in Periods 1 and 2 combined.
Arm/Group | Cohort 1: Gefapixant 300 mg/Chronic Cough | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 12 | 12 | 11
Score on a scale
  Day 1 | 28.2 (30.71) | 35.7 (24.32) | 30.9 (27.22) | 20.5 (12.75)
  Day 2 | 25.8 (30.20) | 44.3 (27.43) | 39.8 (28.97) | 35.5 (22.25)

12. Secondary Outcome: Cough Severity in Response to ATP Challenge (Chronic Cough Participants Only)
Description: In response to ATP challenge in Periods 3 and 4, participants with chronic cough completed a VAS at the end of a 4-hour post-dose observation period on Day 1; and at end of 24-hour observation period on Day 2. For both periods, participants were asked to mark on a 100 mm VAS their cough severity between 0 mm (no cough) and 100 mm (worst cough).
Time Frame: At the end of a 4-hour post-dose observation period on Day 1; at the end of a 24-hour observation period on Day 2
Population: All randomized participants with chronic cough who received at least 1 dose of study medication and had at least 1 post-dose secondary endpoint assessment of cough severity in response to ATP challenge
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Cohort 1: Placebo/Chronic Cough: Participants with chronic cough in Cohort 1 who received placebo in Periods 3 and 4 combined
- Cohort 2: Gefapixant 50 mg/Chronic Cough: Participants with chronic cough in Cohort 2 who received gefapixant 50 mg in Periods 3 and 4 combined
- Cohort 2: Placebo/Chronic Cough: Participants with chronic cough in Cohort 2 who received placebo in Periods 3 and 4 combined
Arm/Group | Cohort 1: Gefapixant 300 mg/Chronic Cough | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 12 | 11 | 11
Score on a scale
  Day 1 | 21.5 (27.06) | 32.7 (24.23) | 21.2 (21.04) | 23.5 (16.02)
  Day 2 | 18.9 (18.29) | 36.8 (26.50) | 27.5 (26.78) | 35.5 (24.07)

13. Secondary Outcome: Daytime Cough Frequency in Participants With Chronic Cough Who Underwent Capsaicin Challenge
Description: Daily cough frequency monitoring was performed in participants with chronic cough, who were attached to a digital sound recorder with 2 microphones (a lapel air microphone attached to the participant's clothing and an adhesive chest wall microphone attached to the skin at the top of the sternum). Participants wore the sound recorder from the start of capsaicin challenge to bedtime on Day 1 in Periods 1 and 2. The resulting recording was processed by software which cut out the majority of speech and background noise but retained cough sounds. The investigator listened to the recording and documented the number of coughs per hour.
Time Frame: From start of challenge (2 hours post-dose) to bedtime; up to 12 hours
Population: All randomized participants with chronic cough who received at least 1 dose of study medication and had at least 1 post-dose secondary endpoint assessment of daytime cough frequency in response to capsaicin challenge
Measure: Mean (Standard Deviation); unit: coughs/hour
Groups:
- Cohort 2: Placebo/Chronic Cough: Participants with chronic cough in Cohort 2 who received single doses of placebo in treatment Periods 1 and 2 combined
Arm/Group | Cohort 1: Gefapixant 300 mg/Chronic Cough | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 12 | 12 | 12
coughs/hour | 13.7 (13.85) | 19.1 (16.76) | 15.5 (16.92) | 20.3 (13.27)

14. Secondary Outcome: Daytime Cough Frequency in Participants With Chronic Cough Who Underwent ATP Challenge
Description: Daily cough frequency monitoring was performed in participants with chronic cough, who were attached to a digital sound recorder with 2 microphones (a lapel air microphone attached to the participant's clothing and an adhesive chest wall microphone attached to the skin at the top of the sternum). Participants wore the sound recorder from the start of ATP challenge to bedtime on Day 1 in Periods 3 and 4. The resulting recording was processed by software which cut out the majority of speech and background noise but retained cough sounds. The investigator listened to the recording and documented the number of coughs per hour.
Time Frame: From start of challenge (2 hours post-dose) to bedtime; up to 12 hours
Population: All treated participants with chronic cough who had at least 1 post-dose secondary endpoint assessment of daytime cough frequency in response to ATP challenge
Measure: Mean (Standard Deviation); unit: coughs/hour
Arm/Group | Cohort 1: Gefapixant 300 mg/Chronic Cough | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
Number analyzed (Participants) | 12 | 12 | 11 | 11
coughs/hour | 10.3 (11.65) | 22.3 (15.48) | 15.6 (17.31) | 26.4 (16.75)

15. Secondary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to Day 41
Population: All randomized participants who received at least 1 dose of study medication
Measure: Number; unit: Percentage of participants
Groups:
- Cohort 1: Gefapixant 300 mg/Healthy: Healthy participants in Cohort 1 who received singles doses of gefapixant 300 mg
- Cohort 1: Placebo/Healthy: Healthy participants in Cohort 1 who received single doses of placebo
- Cohort 1: Gefapixant 300 mg/Chronic Cough: Participants with chronic cough in Cohort 1 who received single doses of gefapixant 300 mg
- Cohort 1: Placebo/Chronic Cough: Participants with chronic cough in Cohort 1 who received single doses of placebo
- Cohort 2: Gefapixant 50 mg/Healthy: Healthy participants in Cohort 2 who received single doses of gefapixant 50 mg
- Cohort 2: Placebo/Healthy: Healthy participants in Cohort 2 who received single doses of placebo
- Cohort 2: Gefapixant 50 mg/Chronic Cough: Participants with chronic cough in Cohort 2 who received single doses of gefapixant 50 mg
- Cohort 2: Placebo/Chronic Cough: Participants with chronic cough in Cohort 2 who received single doses of placebo
Arm/Group | Cohort 1: Gefapixant 300 mg/Healthy | Cohort 1: Placebo/Healthy | Cohort 1: Gefapixant 300 mg/Chronic Cough | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Healthy | Cohort 2: Placebo/Healthy | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12 | 12 | 12 | 11
Percentage of participants | 100.0 | 35.7 | 100.0 | 58.3 | 75.0 | 33.3 | 50.0 | 27.3

16. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an Adverse Event
Description: as for outcome 15
Time Frame: Up to Day 24
Population: All randomized participants who received at least 1 dose of study medication
Measure: Number; unit: Percentage of participants
Groups:
- Cohort 1: Gefapixant 300 mg/Healthy: Healthy participants in Cohort 1 who received single doses of gefapixant 300 mg
- Cohort 1: Gefapixant 300 mg/Chronic Cough: Participants with chronic cough in Cohort 1 who received singles doses of gefapixant 300 mg
Arm/Group | Cohort 1: Gefapixant 300 mg/Healthy | Cohort 1: Placebo/Healthy | Cohort 1: Gefapixant 300 mg/Chronic Cough | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Healthy | Cohort 2: Placebo/Healthy | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
Number analyzed (Participants) | 14 | 14 | 12 | 12 | 12 | 12 | 12 | 11
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Up to Day 41
Description: All randomized participants who received at least 1 dose of study medication.
Arm/Group | Cohort 1: Gefapixant 300 mg/Healthy | Cohort 1: Placebo/Healthy | Cohort 1: Gefapixant 300 mg/Chronic Cough | Cohort 1: Placebo/Chronic Cough | Cohort 2: Gefapixant 50 mg/Healthy | Cohort 2: Placebo/Healthy | Cohort 2: Gefapixant 50 mg/Chronic Cough | Cohort 2: Placebo/Chronic Cough
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 14/14 | 5/14 | 12/12 | 7/12 | 9/12 | 4/12 | 6/12 | 3/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Gefapixant 300 mg/Healthy (N=14) | Cohort 1: Placebo/Healthy (N=14) | Cohort 1: Gefapixant 300 mg/Chronic Cough (N=12) | Cohort 1: Placebo/Chronic Cough (N=12) | Cohort 2: Gefapixant 50 mg/Healthy (N=12) | Cohort 2: Placebo/Healthy (N=12) | Cohort 2: Gefapixant 50 mg/Chronic Cough (N=12) | Cohort 2: Placebo/Chronic Cough (N=11)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth deposit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 13 (20) | 1 (1) | 9 (15) | 1 (1) | 4 (5) | 0 (0) | 3 (5) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 5 (5) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Hypogeusia (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
VIIth Nerve Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No data collected as part of this study will be utilized in any written work, including publications, without the written consent of Sponsor. These obligations of confidentiality and non-use shall in no way diminish such obligations as set forth in the Confidentiality Agreement between the Sponsor and the Investigator(s).